CLINICAL TRIAL: NCT02431767
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of PENNVAX®-GP (Gag, Pol, Env) DNA Vaccine and IL-12 Plasmid, Delivered Via Intradermal or Intramuscular Electroporation in Healthy, HIV-Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of PENNVAX®-GP DNA Vaccine and IL-12 Plasmid, Delivered Via Intradermal or Intramuscular Electroporation in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 098; 11890 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1: Treatment (Experimental): Participants will receive the PENNVAX®-GP vaccine 0.6 mg admixed with IL-12 DNA 0.2 mg to be administered as 0.1 mL by intradermal (ID) injection over either deltoid at Months 0, 1, 3, and 6 using the CELLECTRA® 3P EP system.
  Interventions: Biological: PENNVAX®-GP HIV-1 DNA vaccine; Biological: Interleukin-12 (IL-12) DNA adjuvant
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo to be administered as 0.1 mL ID over either deltoid at Months 0, 1, 3, and 6 using the CELLECTRA® 3P EP system.
  Interventions: Biological: Placebo
- Group 2: Treatment (Experimental): Participants will receive the PENNVAX®-GP vaccine 0.8 mg to be administered as 0.1 mL ID over their left and right deltoids (unless medically contraindicated) at Months 0, 1, 3, and 6 using the CELLECTRA® 3P EP system.
  Interventions: Biological: PENNVAX®-GP HIV-1 DNA vaccine
- Group 2: Placebo (Placebo Comparator): Participants will receive placebo to be administered as 0.1 mL ID over their left and right deltoids (unless medically contraindicated) at Months 0, 1, 3, and 6 using the CELLECTRA® 3P EP system.
  Interventions: Biological: Placebo
- Group 3: Treatment (Experimental): Participants will receive the PENNVAX®-GP vaccine 0.8 mg admixed with IL-12 DNA 0.2 mg to be administered as 0.1 mL ID over their left and right deltoids (unless medically contraindicated) at Months 0, 1, 3, and 6 using the CELLECTRA® 3P EP system.
  Interventions: Biological: PENNVAX®-GP HIV-1 DNA vaccine; Biological: Interleukin-12 (IL-12) DNA adjuvant
- Group 3: Placebo (Placebo Comparator): Participants will receive placebo to be administered as 0.1 mL ID over their left and right deltoids (unless medically contraindicated) at Months 0, 1, 3, and 6 using the CELLECTRA® 3P EP system.
  Interventions: Biological: Placebo
- Group 4: Treatment (Experimental): Participants will receive the PENNVAX®-GP vaccine 8 mg admixed with IL-12 DNA 1 mg to be administered as 1 mL intramuscular (IM) injection in either deltoid at Months 0, 1, 3, and 6 using the CELLECTRA® 5P EP system.
  Interventions: Biological: PENNVAX®-GP HIV-1 DNA vaccine; Biological: Interleukin-12 (IL-12) DNA adjuvant
- Group 4: Placebo (Placebo Comparator): Participants will receive placebo to be administered as 1 mL IM in either deltoid at Months 0, 1, 3, and 6 using the CELLECTRA® 5P EP system.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PENNVAX®-GP HIV-1 DNA vaccine — Administered by intradermal (ID) injection in Groups 1, 2, and 3; administered by intramuscular (IM) injection in Group 4.
  Arms: Group 1: Treatment; Group 2: Treatment; Group 3: Treatment; Group 4: Treatment
Biological: Interleukin-12 (IL-12) DNA adjuvant — Administered by intradermal (ID) injection in Groups 1, 2, and 3; administered by intramuscular (IM) injection in Group 4.
  Arms: Group 1: Treatment; Group 3: Treatment; Group 4: Treatment
Biological: Placebo — Sterile Water for Injection, USP. Administered by intradermal (ID) injection in Groups 1, 2, and 3; administered by intramuscular (IM) injection in Group 4.
  Arms: Group 1: Placebo; Group 2: Placebo; Group 3: Placebo; Group 4: Placebo

SUMMARY:
The study will evaluate the safety and tolerability of the PENNVAX®-GP HIV-1 DNA vaccine and interleukin 12 (IL-12) DNA adjuvant, given by intradermal (ID) or intramuscular (IM) injection with electroporation (EP), in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of the PENNVAX®-GP HIV-1 DNA vaccine and IL-12 DNA adjuvant, given by intradermal (ID) or intramuscular (IM) injection with electroporation (EP), in healthy, HIV-uninfected adults. All study injections will be given using an EP device, which uses an electric pulse to briefly open tiny pores in the cells. Researchers will evaluate whether EP increases the immune response to the vaccine.

The study will enroll participants in four groups. Within each group, participants will be randomly assigned to receive the PENNVAX®-GP DNA vaccine/IL-12 DNA adjuvant or placebo. Each group will receive different doses of the vaccine. Enrollment will begin with Group 1, which will receive a low dose of the vaccine and adjuvant. Study staff will review safety data from Group 1 before enrolling people in Groups 2, 3, and 4 at higher doses. Participants in all groups will receive injections at study entry (Day 0) and Months 1, 3, and 6. At each injection visit, participants in Groups 1 and 4 will receive injections in one arm, and participants in Groups 2 and 3 will receive injections in both arms. Groups 1, 2, and 3 will receive ID injections, and Group 4 will receive IM injections.

Participants will attend study visits at Day 0, Week 2, and Months 1, 1.5, 3, 3.5, 6, 6.5, 9, and 12. Visits will include physical examinations, urine collection, blood collection, HIV and risk reduction counseling, and assessments and questionnaires. Some participants may have photographs taken of the injection site (this is optional). Study staff will contact participants at Month 18 for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria:

* Age of 18 to 55 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit

Laboratory Inclusion Values:

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female, greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal; creatine phosphokinase (CPK) less than or equal to 2.0 times the institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: participants must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status:

* Participants who were born female: negative serum or urine beta human chorionic gonadotropin pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* A participant who was born female must:

  * Agree to consistently use effective contraception (see Appendix B of the protocol) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. More information on this criterion is available in the protocol.
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 098 study
* Pregnant or breastfeeding
* Subcutaneous contraceptive device

Vaccines and Other Injections:

* HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the HVTN 098 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For participants who have received control/placebo in an experimental vaccine trial, the HVTN 098 PSRT will determine eligibility on a case-by-case basis. For participants who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 098 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System:

* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] low-dose inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.
* Serious adverse reactions to vaccines, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency

Clinically Significant Medical Conditions:

* History or presence of keloid scar formation or hypertrophic scar
* Presence of implanted electronic medical device (e.g., pacemaker, implantable cardioverter defibrillator)
* Presence of surgical or traumatic metal implant in the upper arm and/or upper torso
* History of cardiac arrhythmia (e.g., supraventricular tachycardia, atrial fibrillation, or frequent ectopy)
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion is available in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent. For example:

  * Tattoo overlying the injection site
  * Skin conditions at the injection site
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis prophylaxis or therapy
* Asthma exclusion criteria:

  * Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program Expert Panel report).
  * Exclude a participant who:
  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following: 1) Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids; 2) Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06-08 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Frequency of reactogenicity signs and symptoms | Measured through Month 18
Severity of reactogenicity signs and symptoms | Measured through Month 18
Magnitude of local injection/EP site pain as measured by a visual analog scale (VAS) | Measured through Month 18
Frequency of adverse events (AEs) | Measured through Month 18
  Categorized by MedDRA body system, MedDRA preferred term, severity, and assessed relationship to study products.
Measurement of white blood cells | Measured through Month 12
Measurement of neutrophils | Measured through Month 12
Measurement of lymphocytes | Measured through Month 12
Measurement of hemoglobin | Measured through Month 12
Measurement of alkaline phosphatase | Measured through Month 12
Measurement of platelets | Measured through Month 12
Measurement of alanine aminotransferase (ALT) | Measured through Month 12
Measurement of aspartate aminotransferase (AST) | Measured through Month 12
Measurement of creatinine | Measured through Month 12
Measurement of creatine phosphokinase (CPK) | Measured through Month 12
Number of participants with early discontinuation of vaccinations | Measured through Month 12
Distribution of responses to questions regarding acceptability of study injection procedures | Measured through Month 12

SECONDARY OUTCOMES:
Response rate of CD4+ T-cell responses measured by flow cytometry, to HIV-1-specific peptide pools representing gag, pol, env following the third and fourth vaccinations | Measured through Month 12
Response rate of CD8+ T-cell responses measured by flow cytometry, to HIV-1-specific peptide pools representing gag, pol, env following the third and fourth vaccinations | Measured through Month 12
Frequency and magnitude of HIV-1 specific binding antibody (Ab) responses as assessed by multiplex assay following the third and fourth vaccinations | Measured through Month 12
Neutralizing antibody magnitude and breadth against tier 1 and, if applicable, tier 2 HIV-1 isolates as assessed by area under the magnitude-breadth curves following the third and fourth vaccinations | Measured through Month 12
B-cell response rate and magnitude measured by B-cell enzyme-linked immunospot (ELISpot) to quantify Env-specific antibody producing B cells following the third and fourth vaccinations | Measured through Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Srilatha Edupuganti, Study Chair — Emory University
Locations (4):
- United States (4):
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Derived] De Rosa SC, Edupuganti S, Huang Y, Han X, Elizaga M, Swann E, Polakowski L, Kalams SA, Keefer MC, Maenza J, Lu Y, Wise MC, Yan J, Morrow MP, Khan AS, Boyer JD, Humeau L, White S, Pensiero M, Sardesai NY, Bagarazzi ML, Weiner DB, Ferrari G, Tomaras GD, Montefiori DC, Corey L, McElrath MJ; HIV Vaccine Trials Network (HVTN) 098 Study Team. Robust antibody and cellular responses induced by DNA-only vaccination for HIV. JCI Insight. 2020 Jul 9;5(13):e137079. doi: 10.1172/jci.insight.137079. PMID 32437332